CLINICAL TRIAL: NCT01126073
Title: A Double Blind, Randomized Study to Compare Influence of Niacin/Laropiprant on Functional and Morphological Characteristics of Arterial Wall and Parameters of Inflammation in Subjects With Coronary Heart Disease Already Treated With a Statin
Brief Title: Niacin/Laropiprant and Endothelial Function
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Miran Sebestjen, assist. prof. Mirasn Sebestjen Mdf, PhD, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 127-00
Record Dates: First submitted 2010-05-07; First posted 2010-05-19 (Estimated); Last update posted 2011-10-06 (Estimated); Status verified 2011-10

CONDITIONS: Coronary Heart Disease
Keywords: niacin/laropiprant; endothelial function
MeSH Terms: conditions — Coronary Disease | interventions — Niacin; MK-0524

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Niacin/Laropiprant 2000mg/40 mg (Active Comparator): After two weeks patients, who have already been on a stable dose of a statin for at least 6 weeks, will be randomized in the ratio 1:1 to either receive ER niacin/laropiprant or placebo in addition to the statin therapy. Patients in the ER niacin/laropiprant group will receive 1000mg/20 mg tablet for 4 weeks, after that the dose will be increased to 2000mg/40mg tablet. The intention is that all patients receive 2000 mg/40mg dose for the rest of the study period, but should they be intolerant to the higher dose, the maximum tolerated dose will be used.
  Interventions: Drug: Niacin/laropiprant

INTERVENTIONS:
Drug: Niacin/laropiprant — After two weeks patients, who have already been on a stable dose of a statin for at least 6 weeks, willer receive ER niacin/laropiprant in addition to the statin therapy. Patients will receive ER niacin/laropiprant 1000mg/20 mg tablet for 4 weeks, after that the dose will be increased to 2000mg/40mg tablet. The intention is that all patients receive 2000 mg/40mg dose for the rest of the study period, but should they be intolerant to the higher dose, the maximum tolerated dose will be used.
  Arms: Niacin/Laropiprant 2000mg/40 mg
Drug: Placebo — After two weeks patients, who have already been on a stable dose of a statin for at least 6 weeks, will receive placebo in addition to the statin therapy. Patients will receive 1 tablet for 4 weeks, after that the dose will be increased to 2 tablets for the rest of the study period.
  Arms: placebo

SUMMARY:
Primary objective:

To evaluate the impact of 12 weeks' administration of extended release niacin/laropiprant (ERN/LRPT) compared to placebo added to statin therapy on endothelial dependant dilatation of the arterial wall assessed by brachial vasoreactivity in stable coronary heart disease (CHD) patients.

Secondary objective:

To evaluate the impact of 12 weeks' administration of extended release niacin/laropiprant (ERN/LRPT) compared to placebo added to statin therapy on serum lipids and the parameters of inflammation in stable coronary heart disease (CHD) patients.

CHD-coronary heart disease ER-extended release

DETAILED DESCRIPTION:
Endothelial dysfunction can be regarded as a syndrome which exhibits systemic manifestations and is detectable prior to obvious intimal lesions which are considered to be important factors in the pathogenesis of atherosclerosis and its complications. Endothelial function is determined by the integrated index of all atherogenic and atheroprotective factors present in an individual, including known, as well as yet unknown variables and genetic predispositions. Should the hypothesis of endothelial dysfunction reflecting a vascular phenotype prone to atherogenesis be true, endothelial function could then serve as a marker of an inherent atherosclerotic risk. Dysfunction of either the coronary or peripheral vascular endothelium can be considered an independent predictor of cardiovascular events, offering valuable prognostic information additional to that derived from conventional risk factor assessment. Interventions, such as risk factor modification and treatment with various drugs, including statins and angiotensin-converting enzyme inhibitors, have shown to improve endothelial function.

Endothelial dependant vasomotion has been used as a clinical endpoint for assessment of endothelial function. Testing involves pharmacological and/or physiological stimulation of endothelial release of NO and other vasoactive compounds, and often a comparison of vascular responses to endothelium-independent dilators such as nitroglycerine. Determination of local NO bioavailability not only reflects its influence on vascular tone, but also the other important functions of this molecule, which include thromboregulation, cell adhesion, and proliferation

A non-invasive technique has been developed to evaluate endothelium-dependent, brachial artery FMD. Endothelium of the brachial artery is provoked to release nitric oxide (NO) by the pressure created by inflated sphygmomanometer cuff placed on the forearm distal to the brachial artery and its subsequent release 4-5 minutes later.FMD occurs predominantly as a result of local endothelial release of NO and it can be imaged and quantitated as an index of vasomotor function. The advantages of this high-frequency ultrasonographic imaging of the brachial artery are two-fold: it is non-invasive and it allows repeated measurements.

Large prospective epidemiological studies have demonstrated an inverse correlation of high density lipoprotein cholesterol (HDL-C) and the risk of cardiovascular events. Although the atheroprotective effects of HDL have mainly been attributed to its function in reverse cholesterol transport, lately numerous beneficial effects of HDL such as the improvement of endothelial function, anti-inflammatory, anti-thrombotic, antioxidative effects and the stimulation of endothelial regeneration have been identified. Consequently, therapeutic elevation of HDL become more and more important goal of the treatment of patients with coronary artery disease (CAD). Warnholtz et al recently demonstrated that extended-release (ER) niacin 1000 mg daily significantly improved endothelial function in CAD patients with low HDL-C, but not in normal HDL-C. The biggest obstacle for niacin therapy is flushing which makes many patients non compliant to the prescribed medication.

Tredaptive TM [(ERN/LRPT); Merck & Co., Inc, Whitehouse Station, NJ, USA)] is a combination tablet containing 1 g of extended release niacin (ERN) and 20 mg of laropiprant, highly selective PGD2-receptor (DP1) antagonist, which offers improved tolerability, supporting a simplified 1-2 g dosing paradigm and improved compliance.

Statins and niacin have been shown to improve endothelial function in CAD patients, however, the question whether niacin improves endothelial function in statin treated patients still remains open. What would be the time needed to show an effect is also not known, but based on the recent publication by Warholtz it seems that 12 weeks should be sufficient.

This study would prospectively test influence of the higher dose of ER-niacin (2000mg) than used in the latest publications (1000 mg) in addition to laropiprant (40mg) in the CHD patients with low HDL-C, the subgroup which in the recent publication by Warhnoltz seem to have benefited from the treatment with niacin.

ELIGIBILITY:
Inclusion Criteria:

* Age 35-55
* Confirmed CHD (post MI patients, coronarography and/or cycloergometer)
* Already treated for dyslipidemia with a statin and reaching ESC LDL target
* HDL-C <1.1 mmol/l, TG > 1,7 mmol/l and LDL < 2,6 mmol/L
* Will be enrolled into the trial

Exclusion Criteria:

* 3x increase of liver enzyme tests or CK
* Severe renal insufficiency - creatinin >200 mmol/l
* Acute disease within 6 weeks prior to inclusion
* Hypersensitivity to nicotinic acid
* Other cardiac medication stable for at least 4 weeks prior to enrollment
* Acute MI, CABG, PCI within past 3 months
* Congestive heart failure (CHF) _ NYHA 2
* Ejection fraction < 40% measured within the past 6 months
* Malignancy
* HIV infection or immunodeficiency state
* Stable dose of statin < 6 weeks
* Diabetes mellitus type 1
* Diabetes mellitus type 2 with HbA1C > 7%
* Hypo/hyper thyroidism
* Alcohol or drug abuse

Ages: 35 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-09; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
To evaluate the impact of 12 weeks' administration of extended release niacin/laropiprant (ERN/LRPT) compared to placebo added to statin therapy on endothelial dependant dilatation of the arterial wall assessed by brachial vasoreactivity | 12 weeks
  Ultrasound measurement of endothelial dependent brachial artery dilation before and after treatment will be performed in all patients.

CONTACTS AND LOCATIONS:
Locations (1):
- UMC Ljubljana, Ljubljana, Slovenia